CLINICAL TRIAL: NCT04381208
Title: Datos de la Historia clínica y Del Examen físico y neurológico Que Orientan al diagnóstico de Dolor Originario en la articulación sacroilíaca
Brief Title: Medical Record, Physical and Neurological Data That Orient to the Diagnosis of Sacroiliac Joint Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Collaborators: Hospital General Universitario de Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: 19-04-2019
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-04

CONDITIONS: Sacroiliac Joint Somatic Dysfunction; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sacroiliac joint pain: Patients diagnosed with sacroiliac joint pain on the basis of history, physical examination and diagnostic sacroiliac joint block
  Interventions: Diagnostic Test: Complete clinical examination
- Lumbar pain: Patients diagnosed with other chronic lumbar pathologies on the basis of history, physical examination and radiographic studies
  Interventions: Diagnostic Test: Complete clinical examination

INTERVENTIONS:
Diagnostic Test: Complete clinical examination — Medical history-taking, physical examination with provocative maneuvers, radiographic imaging (if relevant), and sacroiliac joint block (if indicated), facet joint block (if indicated)

SUMMARY:
There are many patients coming daily to our office with the complaint of chronic lumbosacral pain radiating or not to the legs that need a proper diagnosis before any treatment is decided. The diagnosis, based mostly on radiological exams, carries a risk of failure to diagnose the sacroiliac joint as the cause of the pain. The study proposes that a quick interrogatory followed by a physical exam with the adequate provocative testing can raise the suspicion of the diagnosis that the pain is originating from the sacroiliac joint. Thereafter, a diagnostic sacroiliac joint block can be performed. The study aims to correlate findings from patient history and physical examination with eventual diagnosis.

DETAILED DESCRIPTION:
This is a prospective cohort study of patients seeking care for chronic low back pain. All patients will undergo a detailed history and physical examination, followed by other indicated diagnostic testing. The analysis will correlate findings from patient history and physical examination testing with the eventual diagnosis. The goal of the study is to identify key historical and physical examination criteria that raise the suspicion for sacroiliac joint pain, which is commonly underdiagnosed. Failure to diagnose a health condition could lead to inappropriate surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient being evaluated in clinic for chronic low back or buttocks pain with or without radiation to the legs

Exclusion Criteria:

* Patient has already undergone surgery for the condition of interest
* Inflammatory condition
* Active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being evaluated in the clinic for chronic low back pain or buttocks pain with or without radiation to the legs.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2019-04-19 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Final diagnosis | 1-2 months
  Number of participants diagnosed with each condition of interest

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vanaclocha V, Jorda-Gomez P, Saiz-Sapena N, Vanaclocha L, Kennedy J. Diagnostic accuracy of clinical examination to distinguish sacroiliac joint pain as a cause of chronic low back pain. Br J Neurosurg. 2024 Dec 10:1-8. doi: 10.1080/02688697.2024.2433492. Online ahead of print. PMID 39654480